CLINICAL TRIAL: NCT04616937
Title: The Role of the Microbiota-gut-brain Axis in Brain Development and Mental Health: Behavioural
Brief Title: Prebiotics and Mental Health: Behavioural
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Surrey (Other)
Collaborators: FrieslandCampina (Industry)
Responsible Party: Principal Investigator, Katherin Cohen-Kadosh, Principal Investigator, University of Surrey
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: PrebioticStudy
Record Dates: First submitted 2020-10-28; First posted 2020-11-05 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Emotion Regulation; Anxiety
MeSH Terms: conditions — Emotional Regulation; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Galacto-oligosaccharides (GOS) Group (Active Comparator): Daily dose of GOS over 4 weeks
  Interventions: Dietary Supplement: GOS
- Placebo group (Placebo Comparator): Daily dose of maltodextrin over 4 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: GOS — Prebiotic
  Arms: Galacto-oligosaccharides (GOS) Group
Dietary Supplement: Placebo — Placebo
  Arms: Placebo group

SUMMARY:
A behavioural study of the microbiota-gut-brain axis in brain development and mental health

DETAILED DESCRIPTION:
Research suggests that modifying microbial ecology therapeutically via the intake of so-called 'psychobiotics' could help reduce stress responses and symptoms of anxiety and depression (Burnet & Cowen, 2013; Dinan, Stanton, & Cryan, 2013; Tang, Reddy, & Saier, 2014). The term psychobiotics refers to both, beneficial gut bacteria (probiotics), as well as prebiotics, which enhance the growth of beneficial gut bacteria (Sarkar et al., 2016). In a recent study, Schmidt and colleagues explored the effects of prebiotics on the secretion of the stress hormone cortisol and emotional processing in healthy volunteers (Schmidt et al., 2015). They found that cortical awakening response was significantly lower after BimunoÒ-galacto-oligosaccharides (Bimuno) intake over 4 weeks compared with placebo. Moreover, participants exhibited decreased attentional vigilance to negative information in a dot-probe task. Given that anxious people show increased biases towards negative information (Bar-Haim, Lamy, Pergamin, Bakermans-Kranenburg, & van, 2007), this suggests that prebiotic intake may be useful in modifying anxiety-related cognitive mechanisms.

These findings will be extended to a sample of late adolescents in order to investigate how prebiotic intake for 4 weeks affects cognitive functioning, psychological well-being and gut microbiota a sample of 60 undergraduate students (aged 18-25 years).

At time 1 (pre-assessment), participants in both groups will undergo comprehensive behavioural and psychological testing to establish baseline measures of cognitive functioning and psychological well-being (such as anxiety levels) and asked to collect a stool sample at home for 16s rRNA sequencing of the microbiome. Group 1 will then receive a daily dosage of a galactooligosaccharide (GOS) prebiotic over 4 weeks, whereas group 2 will receive a placebo over the same period. At time 2 (post-assessment), both groups will again undergo cognitive and psychological testing and stool sampling.

Hypothesis: It is predicted that the treatment group (GOS) will show improvements in behavioural indices of emotion regulation (e.g. dot probe task) and in self reported psychological measures related to emotion regulation (e.g. anxiety) in comparison to the placebo group. Changes/differences in gut microbiome samples will be explored.

ELIGIBILITY:
Inclusion Criteria:

* Females
* Aged between 18-25

Exclusion Criteria:

* Clinical levels of anxiety and/ or co-morbid diagnoses (e.g. depression)
* Current or previous neurological disorders
* Current or previous psychiatric disorders
* Current or previous gastrointestinal disorders
* Current or previous endocrine disorders
* Antibiotic use 3 months prior to the study
* Regular use of pre- and probiotics, including 3 months prior to the study
* Vegan diets
* BMI >30

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 64 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Behavioural indices of emotion regulation | 4 weeks
  Changes in performance on dot-probe task measured as attentional bias to emotional stimuli in milliseconds in the prebiotic group compared to placebo. Increased attentional bias to positive stimuli and/or decreased attentional bias to negative stimuli is the desired outcome.
Changes in self reported indices of anxiety. | 4 weeks
  Changes in self reported anxiety as measured by the Trait Anxiety subscale of the State-Trait Anxiety Inventory (Spielberger, 1978) in the prebiotic group compared to placebo group. For this inventory, a lower overall score is the desired outcome.
Changes in self reported indices of anxiety 2. | 4 weeks
  Changes in self reported anxiety as measured by the State Anxiety subscale of the State-Trait Anxiety Inventory (Spielberger, 1978) in the prebiotic group compared to placebo group. For this inventory, a lower overall score is the desired outcome.
Changes in self reported indices of anxiety 3. | 4 weeks
  Changes in self reported social anxiety measured by Social Anxiety Scales (La G reca 1999) in the prebiotic group compared to placebo group. For this scale, a lower overall score is the desired outcome.
Changes in self reported emotion regulation (Thought control ability). | 4 weeks
  Changes in the prebiotic group compared to placebo for Thought control ability (Luciano et al 2005). For this questionnaire, a higher overall score is the desired outcome.
Changes in self reported emotion regulation (Emotion regulation strategies). | 4 weeks
  Changes in the prebiotic group compared to placebo for emotion regulation strategies (Gross & John, 2003). For this questionnaire, a higher overall score is the desired outcome.
Changes in self reported mood | 4 weeks
  Changes in the prebiotic group compared to placebo for mood and feelings as measured by the mood and feelings questionnaire (Angold etal., 1995). A lower overall score is the desired outcome.
Changes in self reported depression. | 4 weeks
  Changes in the prebiotic group compared to placebo for depression as measured by the Depression inventory (Beck & Steer, 1984). A lower score is the desired outcome.

SECONDARY OUTCOMES:
Gut microbiota changes | 4 weeks
  Changes in gut microbiome composition in diversity, or in abundance of genera (%) (e.g. Bifidobacterium) from pre to post assessment in prebiotic group compared to placebo OR between prebiotic and placebo groups at post assessment.

OTHER OUTCOMES:
Exploratory: Changes in nutrient intake and food choice | 4 weeks
  Changes in the prebiotic group compared to placebo in nutrient intake and food choice, measured by self-reported food diaries (recorded daily and averaged over 4 days at each testing point) followed by macro- and micronutrient intake analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Surrey, Guildford, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: No